CLINICAL TRIAL: NCT03462433
Title: The Safety and Efficacy of Ruptured Intracranial Aneurysms Embolized Assisted With Stents（SERIAES）.
Brief Title: Treatment of Ruptured Intracranial Aneurysms in China.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Air Force Military Medical University, China (Other); Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, He xuying, Deputy director, department of neurosurgery, southern medical university,Guangzhou, Zhujiang Hospital
Other Study IDs: 2016YFC1300800
Record Dates: First submitted 2018-02-07; First posted 2018-03-12 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Ruptured Intracranial Aneurysms; Unruptured Intracranial Aneurysms; Stent-Assisted Coiling; Non-Stent-Assisted Coiling; Craniotomy Clipping
Keywords: Ruptured Intracranial Aneurysms; Unruptured Intracranial Aneurysms; Prospective cohort study; China

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ruptured intracranial aneurysms is currently a common disease that seriously affects human health and quality of life due to its high morbidity,high mortality and high disability. At present,Ruptured intracranial aneurysms are treated with craniotomy clipping and interventional embolization ,but for ruptured wide-neck intracranial aneurysms, the treatment of craniotomy clipping and coiling embolization are not effective.With the improvement of endovascular treatment materials and techniques, three dimensional coil basket technique, double microcatheter technique, balloon assisted ONYX embolization, simple stent covered aneurysm neck, balloon or stent assisted neck remodeling and coil embolization are used in endovascular treatment of ruptured wide-neck intracranial aneurysms. The treatment methods are different in the intervention effect of ruptured wide-neck intracranial aneurysms, for example, the complications of interventional therapy are lower than craniotomy clipping,but the rate of well functional outcome (mRS ≤2) differed significantly by 3 months follow-up (65.0% vs.75.0%), and there is not standard of treatment in different parts of ruptured wide-neck intracranial aneurysms in our country, the choice of interventional therapy or craniotomy clipping are different in different clinical centers; on the other hand, there are serious problems in the treatment of ruptured wide-neck intracranial aneurysms, because without the relevant guidelines of diagnosis and treatment of ruptured wide-neck intracranial aneurysms, different clinical centers will cause excessive treatment of ruptured wide-neck intracranial aneurysms, not only bring unreasonable utilization of medical resources, but also cause the subject's life and property to be threatened.

The patients with ruptured wide-neck intracranial aneurysms(n=1084) and unruptured intracranial aneurysms(n=300) were included in prospective cohort study, after interventional therapy and craniotomy clipping, setting fixed time for postoperative follow-up, the clinical data and image data were recorded, the safety, efficacy and economic benefits of interventional treatment and craniotomy clipping were compared, providing strategies for the standardized treatment of ruptured wide-neck intracranial aneurysms.

DETAILED DESCRIPTION:
For this study, investigators consulted and hired professionals and experts about data collection, data and methodology, including Data Monitoring Committee, Data Management Committee, Project Academic Committee,Executive Group Project Manager, Project Statistician, Technical Support Center, investigators have a scientific regulations for this project, Project Manager and Executive Group: To ensure the successfully implementation of this project, including charging the daily operations of the study in 6 different research hospitals, organizing the monthly meeting to consider issues raised during the monthly progress of the study, liaising with the steering committee the data management center and statistical center , Data management Committee: To be responsible for setting up and maintain the Electronic Data Capture(EDC) System according to the paper case Report Form (pCRF) designed by principal investigators. To collect and save the pCRF coming from sub-centers. To entry the data into EDC system and keep the same with CRF. To organize training for the investigators about the rules in filling the EDC and pCRF.To determine the frequency of the Data Management Report and to fed it back to the steering committee every three months, Data Monitoring Committee: To determine the frequency of the data monitoring including the source data(Medical records) accuracy, completeness and representativeness comparing the external data(EDC,pCRF） in 12 centers.To report the results after the monitoring back to the steering committee about the missing data, non-reported and other problems about the study. To make a Standard Operation Procedure (SOP) from getting data to using data. Academic Committee: To supervise the academic issues including patient recruitment, protocol deviation, adverse events evaluating. To settle down the question and problem in the process of the study, Project Statistician: We cooperate with the Statisticians of Medical Research & Biometrics center National Center for Cardiovascular Diseases, China ti get the professional statistical report. Technical Support Center: To provide technical support during the process of the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least one imaging methods( CTA/ MRA/DSA ) confirmed ruptured wide-neck intracranial aneurysms (fundus-to-neck ratio < 2 or neck diameter > 4 mm );
2. Stent-Assisted Coiling of un-ruptured intracranial aneurysms, whether have clinical symptoms or no;
3. For multiple aneurysms, regardless of previous treatment, the requirement for treatment interval should >6 months;
4. The subjects age 14 years;
5. subjects or family members agree to sign informed consent.

Exclusion Criteria:

1. Subjects with other intracranial vascular malformations, such as AVM, AVF. Etc;
2. Subjects with malignant tumors in the intracranial or other parts of the body;
3. Fusiform, traumatic, bacterial or dissecting aneurysm;
4. Subjects with severe mental illness unable to communicate when diagnosing disease;
5. The body condition is poor, the survival time is less than 1 year or poor physical condition, cannot tolerate the general anesthesia or aneurysm surgery;
6. Subjects involved in other intracranial aneurysms related clinical research;
7. A patient who received surgical clipping or endovascular treatment at once;
8. Subjects who were not followed up；

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ruptured intracranial aneurysms and un-ruptured intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 1384 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
The safety evaluation of interventional therapy and craniotomy clipping. | 6 months later after operation.
  2.The safety evaluation including the mortality(mRS=6) rate and disability(3<mRS<6) rate of subjects.
The safety evaluation of interventional therapy and craniotomy clipping. | 6 months later after operation.
  The safety evaluation including the mortality(mRS=6) rate of subjects.
Modified Rankin score ( mRS ). | 1 year.
  0. completely silent.
  1. despite symptoms, but not visibly disabled, can complete all regular duties and activities
  2. mild disabilities, not all activities previously possible, but can deal with personal affairs without need of assistance
  3. moderate disability requires some help, but walking does not need assistance
  4. severe disabilities, unable to walk independently, no others can not meet their needs
  5. severely disabled, bedridden, Urine, requiring continuous care and care
  6. mortality.
Raymond classification. | 1 year.
  1. Complete occlusion
  2. Partial occlusion
  3. Recurrence.
The effectiveness evaluation of craniotomy clipping. | 6 months later after operation.
  The effectiveness evaluation including the complete occlusion( Raymond classification=1) rate of aneurysms.
The effectiveness evaluation of interventional treatment. | 6 months later after operation.
  The effectiveness evaluation including the recurrence ( Raymond classification =3) rate of aneurysms.
The effectiveness evaluation of craniotomy clipping. | 6 months later after operation.
  The effectiveness evaluation including the recurrence( Raymond classification=3) rate of aneurysms.

SECONDARY OUTCOMES:
The safety evaluation interventional therapy. | 12 months later after operation.
  The safety evaluation including the mortality( mRS=6)rate and disability(3<mRS<6 ) rate of subjects.
The effectiveness evaluation of interventional treatment. | 12 months later after operation.
  The effectiveness evaluation including the complete occlusion( Raymond classification=1 ) rate of aneurysms.
The success rate of treatment. | 6 months later after operation.
  Angiography revealed total or near total occlusion of aneurysm in 6 months after operation, no recurrence of aneurysm was found. the treatment was considered successful.
The incidence of major adverse events after 3 months of surgery. | 3 months.
The incidence of major adverse events in 3 months and 6 months later after operation. | 3 months and 6 months later after operation.
The incidence of major adverse events in 6 months and 12 months later after operation. | 6 months and 12 months later after operation.
The safety evaluation of craniotomy clipping. | 12 months later after operation.
  The safety evaluation including the mortality( MRS=6 ) rate and disability(3<MRS <6) rate of subjects.
The effectiveness evaluation of interventional treatment. | 12 months later after operation.
  The effectiveness evaluation including the recurrence( Raymond classification=3 ) rate of aneurysms.
The effectiveness evaluation of craniotomy clipping. | 12 months later after operation.
  The effectiveness evaluation including the complete occlusion( Raymond classification=1 ) rate of aneurysms.
The effectiveness evaluation of craniotomy clipping. | 12 months later after operation.
  The effectiveness evaluation including the recurrence( Raymond classification=3) rate of aneurysms.

CONTACTS AND LOCATIONS:
Overall Officials: Xuying He, PH. D, Principal Investigator — Study Principal Investigator Department of Neurosurgery, Southern Medical University, Zhujiang Hospital
Locations (1):
- Southern Medical University, Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
investigators can share the original data 5 years after the study